CLINICAL TRIAL: NCT00575315
Title: HIV-HCV Coinfection: Impact of Immune Dysfunction
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: VCU03488; K23-DK-066578-01
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: HIV Infections; Hepatitis
Keywords: HIV-HCV Coinfection; HIV; Histology
MeSH Terms: conditions — HIV Infections; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sera
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Effective therapy for human immunodeficiency virus (HIV) infection has markedly prolonged survival in infected individuals. As a result, other diseases are now becoming clinically significant. Approximately 30% of HIV infected patients are co-infected with hepatitis C virus (HCV) which is now the leading co-morbid disease in co-infected individuals. The histologic severity and natural history of HCV has been reported to be accelerated in those co-infected with HIV. It is hypothesized that 1) the severity and progression of HCV disease is related to the immune competence of the individual, 2) immune restoration associated with HIV therapy may further accelerate the progression of HCV disease which may explain the marked increase in HCV related morbidity and mortality observed in recent years, and 3) the virologic response to anti-HCV treatment is directly related to the degree of immunologic competence. The specific aims of the proposal are: 1) To obtain, through multi-disciplinary didactic teaching, the necessary skills of clinical research design, data collection, data analysis, and biostatistical methods and 2) To study the impact of HIV disease on HCV, the effect of the immune function and immune restoration during HIV therapy on the natural history of HCV, and the efficacy of HCV treatment in HIV co-infection.

DETAILED DESCRIPTION:
Approximately 30% of HIV infected patients are co-infected with hepatitis C virus (HCV) which is now the leading co-morbid disease in co-infected individuals. The histologic severity and natural history of HCV has been reported to be accelerated in those co-infected with HIV. It is hypothesized that 1) the severity and progression of HCV disease is related to the immune competence of the individual, 2) immune restoration associated with HIV therapy may further accelerate the progression of HCV disease which may explain the marked increase in HCV related morbidity and mortality observed in recent years, and 3) the virologic response to anti-HCV treatment is directly related to the degree of immunologic competence. The specific aims of the proposal are: 1) To obtain, through multi-disciplinary didactic teaching, the necessary skills of clinical research design, data collection, data analysis, and biostatistical methods and 2) To study the impact of HIV disease on HCV, the effect of the immune function and immune restoration during HIV therapy on the natural history of HCV, and the efficacy of HCV treatment in HIV co-infection.

ELIGIBILITY:
Inclusion Criteria:

* HIV antibody positive
* Positive HCV-RNA
* Age > 18 years

Exclusion Criteria:

* Coagulopathy (prothrombin time prolonged > 2 seconds from control)
* Presence of ascites
* Thrombocytopenia (platelet < 70,000)
* Active or recent (within 3 months) opportunistic infection related to HIV
* Advanced HIV disease with life expectancy less than 1 year
* Renal failure
* Hepatitis B surface antigen positive
* Inability to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-HCV Coinfection
Sampling Method: Non-Probability Sample
Enrollment: 634 (Actual)
Dates: Start 2004-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Changes in liver histology | 5 years

SECONDARY OUTCOMES:
Assessing the effect of confounding variables on hepatic fibrosis. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Sterling, MD MSc, Principal Investigator — VCU
Locations (1):
- Virgnia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] Shah AG, Smith PG, Sterling RK. Comparison of FIB-4 and APRI in HIV-HCV coinfected patients with normal and elevated ALT. Dig Dis Sci. 2011 Oct;56(10):3038-44. doi: 10.1007/s10620-011-1710-2. Epub 2011 Apr 28. PMID 21526398
- [Background] Sterling RK, Wegelin JA, Smith PG, Stravitz RT, Luketic VA, Fuchs M, Puri P, Shiffman ML, Contos MA, Mills AS, Sanyal AJ. Similar progression of fibrosis between HIV/HCV-infected and HCV-infected patients: Analysis of paired liver biopsy samples. Clin Gastroenterol Hepatol. 2010 Dec;8(12):1070-6. doi: 10.1016/j.cgh.2010.08.004. Epub 2010 Aug 20. PMID 20728569
- [Background] Sterling RK, Contos MJ, Smith PG, Stravitz RT, Luketic VA, Fuchs M, Shiffman ML, Sanyal AJ. Steatohepatitis: Risk factors and impact on disease severity in human immunodeficiency virus/hepatitis C virus coinfection. Hepatology. 2008 Apr;47(4):1118-27. doi: 10.1002/hep.22134. PMID 18366118
- [Background] Sterling RK, Chiu S, Snider K, Nixon D. The prevalence and risk factors for abnormal liver enzymes in HIV-positive patients without hepatitis B or C coinfections. Dig Dis Sci. 2008 May;53(5):1375-82. doi: 10.1007/s10620-007-9999-6. Epub 2007 Oct 16. PMID 17939038
- [Background] Smith JO, Sterling RK. Hepatitis C and HIV. Curr Gastroenterol Rep. 2007 Mar;9(1):83-90. doi: 10.1007/s11894-008-0025-8. PMID 17335682
- [Background] Sterling RK, Lissen E, Clumeck N, Sola R, Correa MC, Montaner J, S Sulkowski M, Torriani FJ, Dieterich DT, Thomas DL, Messinger D, Nelson M; APRICOT Clinical Investigators. Development of a simple noninvasive index to predict significant fibrosis in patients with HIV/HCV coinfection. Hepatology. 2006 Jun;43(6):1317-25. doi: 10.1002/hep.21178. PMID 16729309
- [Background] Sterling RK, Brown RS Jr, Hofmann CM, Luketic VA, Stravitz RT, Sanyal AJ, Contos MJ, Mills AS, Smith V, Shiffman ML. The spectrum of chronic hepatitis C virus infection in the Virginia Correctional System: development of a strategy for the evaluation and treatment of inmates with HCV. Am J Gastroenterol. 2005 Feb;100(2):313-21. doi: 10.1111/j.1572-0241.2005.40116.x. PMID 15667488
- [Background] Stravitz RT, Shiffman ML, Sanyal AJ, Luketic VA, Sterling RK, Heuman DM, Ashworth A, Mills AS, Contos M, Cotterell AH, Maluf D, Posner MP, Fisher RA. Effects of interferon treatment on liver histology and allograft rejection in patients with recurrent hepatitis C following liver transplantation. Liver Transpl. 2004 Jul;10(7):850-8. doi: 10.1002/lt.20189. PMID 15237368
- [Background] Sterling RK, Wilson MS, Sanyal AJ, Luketic VA, Stravitz RT, Contos MJ, Mills AS, Shiffman ML. Impact of highly active antiretroviral therapy on the spectrum of liver disease in HCV-HIV coinfection. Clin Gastroenterol Hepatol. 2004 May;2(5):432-9. doi: 10.1016/s1542-3565(04)00129-6. PMID 15118983
- [Background] Sterling RK, Contos MJ, Sanyal AJ, Luketic VA, Stravitz RT, Wilson MS, Mills AS, Shiffman ML. The clinical spectrum of hepatitis C virus in HIV coinfection. J Acquir Immune Defic Syndr. 2003 Jan 1;32(1):30-7. doi: 10.1097/00126334-200301010-00005. PMID 12514411